CLINICAL TRIAL: NCT02993939
Title: A Randomized Comparison Between Interscalene Brachial Plexus Block and Combined Infraclavicular Brachial Plexus Block-Suprascapular Nerve Block
Brief Title: Interscalene Block Versus Infraclavicular Block Plus Suprascapular Nerve Block
Acronym: ISBvsICB-SSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, MD Clinical Instructor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 853/16
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Shoulder Injury
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interscalene block (Active Comparator): Ultrasound guided Brachial plexus block injecting 20 ml of levobupivacaine 0,25% plus epinephrine 5 micrograms per ml, in the Interscalene groove.
  Interventions: Procedure: Interscalene block
- Diaphragm-sparing block (Experimental): Ultrasound guided combinated infraclavicular-Suprascapular block of the braquial plexus, injecting 20 ml of levobupivacaine 0,25% plus epinephrine 5 micrograms per ml dorsal to the axillary artery in the infraclavicular fossa plus an Ultrasound guided injection of 10 ml of levobupivacaine 0,25% plus epinephrine 5 micrograms per ml in the suprascapular fossa.
  Interventions: Procedure: Infraclavicular-suprascapular block

INTERVENTIONS:
Procedure: Interscalene block — Ultrasound guided single shot block above the clavicle
  Arms: Interscalene block
Procedure: Infraclavicular-suprascapular block — Combined block of nerves far away from phrenic nerve
  Arms: Diaphragm-sparing block

SUMMARY:
Despite their reliability and efficacy for shoulder surgery analgesia, above clavicle brachial plexus blocks are related with phrenic nerve palsy and diaphragm paralysis that may not be tolerated in patients with chronic pulmonary disease.

This RCT will compare the classic Interscalene block with combined infraclavicular block plus suprascapular nerve block in patients going for arthroscopic shoulder surgery.

Main outcome is static pain in the recovery room measured with NRS. Secondary outcomes are pain at 12 and 24 hrs and incidence of diaphragmatic paralysis.

DETAILED DESCRIPTION:
PATIENT RECRUITMENT

With the approval of the Ethics Committee of Hospital Clinico Universidad de Chile, 40 patients undergoing arthroscopic shoulder surgery will be recruited. Enrollment will be carried out by an investigator not involved in patient care. Patients' confidentiality will be protected.

STUDY PROTOCOL: GENERAL

All blocks will be performed by one of the coauthors and conducted preoperatively in an induction room. Sedation (2 mg midazolam and 50 μg fentanyl) will be provided for patient comfort.

STUDY PROTOCOL: PERFORMANCE OF THE BLOCK

Both study groups will receive an ultrasound-guided superficial cervical plexus block.

In the ICB-SSB group, suprascapular nerve blocks will be carried out using a previously described technique. For infraclavicular brachial plexus blocks, 20 mL of levobupivacaine 0.25% with epinephrine 5 µg/mL will be injected dorsal to the axillary artery, medial to the coracoid process.

In the ISB group, block will carried out using a previously described technique: 20 mL of levobupivacaine 0.25% with epinephrine 5 µg/mL will be deposited under the prevertebral fascial between the C5 and C6 roots.

STUDY PROTOCOL: GENERAL ANESTHESIA

All patients will undergo standardized general anesthesia

STUDY PROTOCOL: POSTOPERATIVE ANALGESIA

In the Recovery Room, all patients will receive acetaminophen (usual dose…) and ketoprofen (usual dose…) as well as patient controlled analgesia (morphine bolus = 1 mg; lockout interval = 8 minutes). On the surgical ward, all subjects will continue to receive acetaminophen (usual dise…), celecoxib (usual dose…) as well and patient controlled analgesia (morphine bolus = 1 mg IV; lockout interval = 8 minutes).

STUDY PROTOCOL: OUTCOME MEASUREMENTS

The primary outcome will be the pain score in the PACU at 30 30 minutes using a sensorimotor composite scale:

Performance time, sensorimotorSensory function, Onset time

The blinded investigator will also assess the presence of hemidiaphragmatic block at 30 minutes. A 2-6 MHz curvilinear US probe (Sonosite M-Turbo, SonoSite Inc, Bothell, WA, USA) and the M-mode will be employed in all subjects; the liver and spleen will serve as acoustic windows on the right and left side, respectively. Patients will be scanned along the anterior axillary line and the US probe, angled cranially

POTENTIAL BENEFITS OF THE STUDY This study will allow us to determine if ICB-SSB constitutes a viable alternative to ISB.

POTENTIAL SIDE EFFECTS OF THE STUDY Participation in this protocol will not put patients at higher risk for complications since ISB and ICB-SSB are commonly used to provide analgesia for shoulder surgery

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 30

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* obstructive or restrictive pulmonary disease (assessed by history and physical examination)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to local anesthetics (LAs)
* pregnancy
* prior surgery in the neck, infraclavicular region or suprascapular fossa
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-28 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Static Pain using numeric scale 0-10 | 30 minutes after arrival to PACU

SECONDARY OUTCOMES:
Static Pain using numeric scale 0-10 | 12 hrs after arrival to PACU
Diaphragm paralysis incidence | 30 minutes after block
Static Pain using numeric scale 0-10 | 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Result] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Result] Martinez J, Sala-Blanch X, Ramos I, Gomar C. Combined infraclavicular plexus block with suprascapular nerve block for humeral head surgery in a patient with respiratory failure: an alternative approach. Anesthesiology. 2003 Mar;98(3):784-5. doi: 10.1097/00000542-200303000-00031. No abstract available. PMID 12606927
- [Result] Tran DQ, Dugani S, Finlayson RJ. A randomized comparison between ultrasound-guided and landmark-based superficial cervical plexus block. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):539-43. doi: 10.1097/AAP.0b013e3181faa11c. PMID 20975470
- [Result] Chan CW, Peng PW. Suprascapular nerve block: a narrative review. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):358-73. doi: 10.1097/AAP.0b013e3182204ec0. PMID 21654552
- [Result] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654
- [Result] Spence BC, Beach ML, Gallagher JD, Sites BD. Ultrasound-guided interscalene blocks: understanding where to inject the local anaesthetic. Anaesthesia. 2011 Jun;66(6):509-14. doi: 10.1111/j.1365-2044.2011.06712.x. PMID 21568985
- [Result] Flohr-Madsen S, Ytrebo LM, Valen K, Wilsgaard T, Klaastad O. A randomised placebo-controlled trial examining the effect on hand supination after the addition of a suprascapular nerve block to infraclavicular brachial plexus blockade. Anaesthesia. 2016 Aug;71(8):938-47. doi: 10.1111/anae.13504. PMID 27396247
- [Result] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304
- [Result] Dhir S, Sondekoppam RV, Sharma R, Ganapathy S, Athwal GS. A Comparison of Combined Suprascapular and Axillary Nerve Blocks to Interscalene Nerve Block for Analgesia in Arthroscopic Shoulder Surgery: An Equivalence Study. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):564-71. doi: 10.1097/AAP.0000000000000436. PMID 27380105
- [Derived] Aliste J, Bravo D, Finlayson RJ, Tran DQ. A randomized comparison between interscalene and combined infraclavicular-suprascapular blocks for arthroscopic shoulder surgery. Can J Anaesth. 2018 Mar;65(3):280-287. doi: 10.1007/s12630-017-1048-0. Epub 2017 Dec 19. PMID 29270914